CLINICAL TRIAL: NCT02354014
Title: A Phase 2, Open-label, Multicenter, Single-arm Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Anti-mycobacterial Activity of TMC207 in Combination With a Background Regimen (BR) of Multidrug Resistant Tuberculosis (MDR-TB) Medications for the Treatment of Children and Adolescents 0 Months to <18 Years of Age Who Have Confirmed or Probable Pulmonary MDR-TB
Brief Title: Pharmacokinetic Study to Evaluate Anti-mycobacterial Activity of TMC207 in Combination With Background Regimen (BR) of Multidrug Resistant Tuberculosis (MDR-TB) Medications for Treatment of Children/Adolescents Pulmonary MDR-TB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR106371; TMC207-TIDP59-C211 (Other: Janssen Research & Development, LLC); 2014-003372-23 (EudraCT Number)
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multidrug-Resistant Tuberculosis
Keywords: Multidrug-Resistant Tuberculosis; Bedaquiline; TMC207
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Bedaquiline (TMC207)/Background Regimen (BR) (Experimental): There will be 4 age-based cohorts. Participants will be enrolled concurrently in Cohorts 1 and 2 followed by sequential enrollment of Cohorts 3, 4. Cohort 1: >= 12 to < 18 years: bedaquiline (TMC207) tablet orally as 400 mg, once daily(qd),for first 2 weeks, followed by bedaquiline (TMC207), 200 mg 3 times per week (tiw) for 22 weeks; Cohort 2: >=5 to <12 years: TMC207 tablet given orally as 200 mg, qd, for first 2 weeks, followed by bedaquiline (TMC207), 100 mg, tiw for 22 weeks. Cohort 3: >=2 to <5 years: TMC207 8 milligram per kilogram (mg/kg) qd for the first 2 weeks, followed by bedaquiline (TMC207) 4 mg/kg tiw for 22 weeks. Cohort 4: 0 months to <2 years: TMC207 doses will be selected as per weight band and age group. bedaquiline (TMC207) will be given in combination with Background Regimen for Multidrug Resistant Tuberculosis (MDR-TB) according to WHO/national tuberculosis program (NTP) guidelines/current standard of care.
  Interventions: Drug: Bedaquiline (TMC207); Drug: Background Regimen (BR)

INTERVENTIONS:
Drug: Bedaquiline (TMC207) — Bedaquiline (TMC207) oral tablet adult formulation (containing 100 mg bedaquiline (TMC207) per tablet) administered as 400 milligram (mg), once daily, for the first 2 weeks, followed by bedaquiline 200 mg 3 times per week with intakes at least 2 days (48 hours) apart for 22 weeks in cohort 1. Cohort 2, 3 and 4 will receive an age appropriate oral tablet formulation containing 20mg bedaquiline . Bedaquiline tablet administered orally as 200 mg, once daily, for the first 2 weeks, followed by bedaquiline 100 mg 3 times per week with intakes at least 2 days (48 hours) apart for 22 weeks in cohort 2. In Cohort 3, dose of bedaquiline 8 mg/kg qd for the first 2 weeks, followed by bedaquiline 4 mg/kg times weekly (TIW) with intakes at least 2 days (48 hours) apart for 22 weeks will be administered. In cohort 4, bedaquiline (TMC207) qd for the first 2 weeks, followed by bedaquiline TIW with intakes at least 2 days (48 hours) apart for 22 weeks.
  Other Names: Bedaquiline
Drug: Background Regimen (BR) — Background Regimen (BR) of Multidrug Resistant Tuberculosis (MDR-TB) medications will be dosed according to World Health Organization (WHO) guidelines, National Tuberculosis Program (NTP) guidelines and current standard of care at the site.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (explores what the body does to the drug), and anti-mycobacterial activity of bedaquiline (TMC207) in children and adolescents (0 months to less than [<] 18 years of age) diagnosed with confirmed or probable pulmonary multidrug resistant tuberculosis (MDR-TB), in combination With a Background Regimen (BR) of MDR-TB Medications.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a boy or girl, aged from birth (0 months) to less than (<) 18 years at screening. Participants in Cohort 4 who are <6 months of age at screening, gestational age at birth had to be greater than or equal to (>=) 37 weeks
* Participant must weigh >3 kilogram (kg) at baseline and be within the 5th and 95th percentiles (inclusive) for the participant's age, based on the World Health Organization (WHO) child growth standards; Body Mass Index (BMI) for age. In Cohorts 3 and 4, weight for height/length may be used instead of BMI for age according to the local standard of care. Per WHO guidance, for Cohort 4, length will be used to calculate the BMI instead of height
* For Cohorts 1 and 2 only: Heterosexually active girls may participate if they are of non-childbearing potential, or if they are using effective birth control methods and are willing to continue practicing birth control methods throughout Multidrug Resistant Tuberculosis (MDR-TB) treatment and for 6 months after stopping TMC207 treatment, or if they are non-heterosexually active or willing to practice sexual abstinence throughout MDR-TB treatment
* For Cohorts 1 and 2 only: Boys who engage in sexual activity that could lead to pregnancy of the female partner must use at minimum a male condom throughout MDR-TB treatment and for 3 months after stopping TMC207 treatment
* Participant must have confirmed or probable (clinically diagnosed or presumed) pulmonary and/or non-severe extrapulmonary MDR-TB, including pre-extensively drug-resistant TB (pre- extensively drug resistant [XDR]-TB) or XDR-TB infection, based on the case definitions of pediatric pulmonary and non-severe extrapulmonary TB as described in the International (WHO) guidelines and in accordance with the local standard of care
* Participants must be starting the initial MDR-TB treatment at baseline or have started an MDR-TB treatment within 12 weeks of baseline and are willing to modify it if necessary to an acceptable MDR-TB regimen for use with TMC207
* Participant must be willing to permanently discontinue RMP from at least 7 days before the baseline visit
* Participant must consent/assent to human Immunodeficiency virus (HIV) testing. If the potential participant is a child aged <2 years, or if the participant is being breastfed or was breastfed within the last 8 weeks before screening, the mother must also consent to HIV testing unless an HIV test was performed within 1 month prior to screening and documentation of HIV status can be provided. When documented HIV-positive status is available prior to screening for participants in Cohort 4, HIV testing is not required

Exclusion Criteria:

* Participant has a clinically significant active medical condition or the presence of any concomitant severe illness or rapidly deteriorating health condition, including immune deficiency (except HIV infection), which in the opinion of the investigator would prevent appropriate participation in the study, or that would make implementation of the protocol or interpretation of the study results difficult, or otherwise make the subject a poor candidate for a clinical study
* Participant is a girl who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 6 months after stopping TMC207 treatment
* Participant has known or presumed forms of extrapulmonary TB, other than: Lymphadenopathy (peripheral nodes or isolated mediastinal mass without significant airway compression); Pleural effusion or pleural fibrotic lesions
* Participant has a significant cardiac arrhythmia that requires medication or a history of risk factors for Torsade de Pointes, example heart failure, hypokalemia, known personal or family history of Long QT Syndrome, and untreated hypothyroidism

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05-03 (Actual); Primary Completion 2027-02-11 (Estimated); Study Completion 2027-02-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | 120 weeks
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Maximum Plasma Concentration (Cmax) | Week 2 and 12
  The Cmax is the maximum plasma concentration.
Time to Reach Maximum Plasma Concentration (Tmax) | Week 2 and 12
  The Tmax is time to reach the maximum plasma concentration.
Minimum Plasma Concentration (Cmin) | Week 2, 12 and 24
  The Cmin is the minimum plasma concentration.
Area Under the Plasma Concentration-time Curve From the Time of Dose Administration up to X Hours (AUCtime-h) | Week 2, 12 and 24
  AUCtime-h is the area under the plasma concentration-time curve from the time of dose administration up to X hours.
Elimination Half-life (t1/2) | Day 1, week 2, 4,6,8,12,16,20,24,28,32,40,48,60,72,84,96,108,120
  Elimination half-life (t [1/2]) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z). Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Area Under the Plasma Concentration-time Curve From the Time of Dose Administration up to 168 Hours [AUC168h] | Week 12 and 24
  AUC168h is the area under the plasma concentration-time curve from the time of dose administration up to 168 Hours.
Volume of Distribution (Vd) | Day 1, week 2, 4,6,8,12,16,20,24,28,32,40,48,60,72,84,96,108,120
  Volume of distribution is calculated as Dose divided by Lambda(z) multiplied by AUC(infinity). The AUC (infinity) is the area under the plasma concentration-time curve from time zero to infinite time.
Apparent Clearance (CL) | Day 1, week 2, 4,6,8,12,16,20,24,28,32,40,48,60,72,84,96,108,120
  Apparent clearance is calculated as Dose/AUC (infinity). The AUC (infinity) is the area under the plasma concentration-time curve from time zero to infinite time.

SECONDARY OUTCOMES:
Percentage of Participants with Favorable Treatment outcome (Sustained Positive Clinical Cure) | Week 24, Week 120 (end of study)
  Sustained Positive Clinical Cure is defined as the percentage of participants with favorable treatment outcome at Week 24 and at study end.
Time to First Confirmed Sputum Culture Conversion, to acid-fast bacilli (AFB) smear conversion, or Other Microbiology Specimen Sample | Baseline (Day 1) up to Week 120
  Culture conversion is defined as 2 consecutive negative cultures in the Mycobacteria Growth Indicator Tube (MGIT) system at least 25 days apart with the last culture within the analysis window, unless a repeat microbiology sample (eg, lymph node biopsy) cannot be obtained. AFB smear conversion is defined as 2 consecutive negative AFB smear at least 25 days apart.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- Hospital Geral da Polana Caniço, Maputo, Mozambique
- Philippines (3):
  - De La Salle Health Sciences Institute- DLSUMC, Dasmariñas
  - Lung Center Of The Philippines, Quezon City
  - Silang Specialists Medical Center, San Vincent Silang
- First Moscow State Medical University n.a. I.M. Sechenov, Moscow, Russia
- South Africa (4):
  - THINK: Tuberculosis & HIV Investigative Network, Durban
  - Sizwe Tropical Diseases Hospital, Johannesburg
  - Wits Health Consortium, Port Elizabeth
  - Desmond Tutu TB Centre, Stellenboch
- Makerere University Lung Institute, Kampala, Uganda
- State Institute Of Phthisiology And Pulmonology N.A. F.G. Yanovskiy Of Ams Ukraine, Kiev, Ukraine